CLINICAL TRIAL: NCT05497674
Title: A Study In Healthy Subjects To Assess The Effects Of Rifampicin Capsules and Probenecid Tablets On The Pharmacokinetic Profile Of Rongliflozin Capsules
Brief Title: Effects of Rifampicin and Probenecid On The Pharmacokinetic Profile Of Rongliflozin In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DJT1116PG-DM-108
Record Dates: First submitted 2022-08-01; First posted 2022-08-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rongliflozin; Rifampin; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rongliflozin and/or rifampicin (Experimental): on Day 1, subjects will receive a single dose administration of rongliflozin, followed by a washout period of 4 days. Starting On Day 5, subjects will administer rifampicin once a day (QD) for 10 consecutive days ( Day 5 to Study Day 14) , comprising of a single dose administration of rongliflozin on Study Day 11.
  Interventions: Drug: Rongliflozin; Drug: Rifampin
- rongliflozin and/or probenecid (Experimental): on Day 1, subjects will receive a single dose administration of rongliflozin, followed by a washout period of 4 days. Probenecid will be administrated twice a day from Day 5 to Day 9, and another single dose administration of rongliflozin on Day 6.
  Interventions: Drug: Rongliflozin; Drug: Probenecid

INTERVENTIONS:
Drug: Rongliflozin — oral administration, single dose on Day 1 and Day 11
  Arms: rongliflozin and/or rifampicin
Drug: Rifampin — QD for 10 days
  Arms: rongliflozin and/or rifampicin
Drug: Rongliflozin — oral administration, single dose on Day 1 and Day 6
  Arms: rongliflozin and/or probenecid
Drug: Probenecid — twice a day, for 5 days
  Arms: rongliflozin and/or probenecid

SUMMARY:
This is a phase I, open-label, fixed-sequence study in healthy Chinese subjects, performed at a single study centre. Cohort A will assess the Pharmacokinetic (PK) profile of rongliflozin when administered alone and the combination with rifampicin; Cohort B will assess the PK profile of rongliflozin when administered alone and combination with probenecid.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial and fully understand the trial content, process and possible adverse reactions;
* Be able to complete the test according to the requirements of the protocol;
* Subjects (including partners) are willing to take effective contraceptive measures from screening to 6 months after the last dose of drug administration;
* Male subjects weigh at least 50 kg and female subjects at least 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), BMI within the range of 18 to 28 kg/m2 ;
* Physical examination and vital signs are both normal or do not have clinical significance.

Exclusion Criteria:

* Smoking more than 5 cigarettes per day;
* Those who are allergic to or have allergies to the test drug;
* have a history of drug or alcohol abuse;
* Blood donation or massive blood loss (>450 mL) within three months prior to screening;
* Difficulty swallowing or any history of digestive system diseases which could affect drug absorption and excretion within 6 months before screening;
* taking any drugs that could alter liver enzyme activity, such as barbiturates, rifampin, etc., within 30 days before screening;
* have taken any prescription, over-the-counter, vitamin product or herbal medicine within 14 days prior to screening;
* Have taken special diets (including dragon fruit, mango, grapefruit, etc.) or exercised strenuously within 2 weeks before screening;
* Take an inhibitor or inducer of glucuronide transferase (UGT), P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP), such as itraconazole, ketoconazole, or dronedarone, within 30 days before screening;
* Significant changes in dietary or exercise habits within 2 weeks prior to screening; Female subjects are breastfeeding or have a positive blood pregnancy result during the screening period;
* During the screening period, the serum uric acid level was >420 µmol/l, or had a history of gout; during the screening period, the estimated glomerular filtration rate (eGFR) was <90 ml/min/1.73m2) or had a history of kidney stones or bladder stones (applicable to Cohort B);
* have a clinically significant laboratory tests or medical history;
* Positive for hepatitis B, hepatitis C, AIDS, syphilis; positive for urine drug test;
* History of urinary tract infection or genital infection before 6 months
* Those who participated in any drug clinical trial and used the experimental drug 3 months ago;
* Subjects with other factors deemed inappropriate by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
rongliflozin: area under the drug-time curve (AUC) ratios of geometric means of rongliflozin+rifampicin relative to rongliflozin alone. | from 0 hour（pre-dose,within 30mins）to 5 days after rongliflozin dosing
  To assess the effect of rifampicin on the AUC of rongliflozin
rongliflozin: The peak concentration (Cmax) ratios of geometric means of rongliflozin+rifampicin relative to rongliflozin alone. | from 0 hour（pre-dose,within 30mins）to 5 days after rongliflozin dosing
  To assess the effect of rifampicin on the Cmax of rongliflozin
rongliflozin: AUC ratios of geometric means of rongliflozin+probenecid relative to rongliflozin alone. | from 0 hour（pre-dose,within 30mins）to 5 days after rongliflozin dosing
  To assess the effect of probenecid on the AUC of rongliflozin
rongliflozin:Cmax ratios of geometric means of rongliflozin+probenecid relative to rongliflozin alone. | from 0 hour（pre-dose,within 30mins）to 5 days after rongliflozin dosing
  To assess the effect of probenecid on the Cmax of rongliflozin

SECONDARY OUTCOMES:
The time to peak (Tmax) of Rongliflozin. | from 0 hour（pre-dose,within 30mins）to 5 days after rongliflozin dosing
  To assess the effect of rifampicin and probenecid on the Tmax of rongliflozin
pharmacology (PD) of rongliflozin: cumulative urine glucose excretion every 24 hours | from 0 hour to 5 days after rongliflozin dosing
  evaluate the cumulative urine glucose excretion every 24 hours after rongliflozin administration.
the number of participants with adverse events (AE) in Cohort A | from screening to 3 days after last dose of rifampicin
  To evaluate the safety and tolerability of single dose of rongliflozin and combination of rifampin
the number of participants with adverse events (AE) in Cohort B | from screening to 3 days after last dose of probenecid
  To evaluate the safety and tolerability of single dose of rongliflozin and combination of probenecid

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: No